CLINICAL TRIAL: NCT04686110
Title: Analysis of Capillary Retinal and Papillary Vascularization in Patients With Amyotrophic Lateral Sclerosis
Brief Title: Analysis of Capillary Retinal and Papillary Vascularization in Patients With Amyotrophic Lateral Sclerosis - CAPISLA
Acronym: CAPISLA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-AO3395-34
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients Amyotrophic Lateral Sclerosis (Other)
  Interventions: Other: angiographic optical coherence tomography
- Control subjects (Other)
  Interventions: Other: angiographic optical coherence tomography

INTERVENTIONS:
Other: angiographic optical coherence tomography — angiographic optical coherence tomography

SUMMARY:
Amyotrophic Lateral Sclerosis, or Charcot's disease, is a neurodegenerative disease affecting motor neurons. The disease affects between 5 and 10 people per 100,000 in the world, nearly 7,000 patients are affected in France. The only therapeutic treatment available to date in France is riluzole, which slows the progression of the disease. Amyotrophic Lateral Sclerosis is the first degenerative disease affecting motor neurons. However, recent evidence suggests that the impairment extends beyond motor neurons alone.

Optical Coherence Tomography analyzes made it possible to highlight ophthalmologic damage in patients with Amyotrophic Lateral Sclerosis, in particular at the macula and papilla, although some results are contradictory.

No angiographic Optical Coherence Tomography analysis has been performed to date in patients with Amyotrophic Lateral Sclerosis. However, in the hypothesis of microvascular involvement participating in the pathophysiology of neurodegeneration in Amyotrophic Lateral Sclerosis, these examinations could provide relevant clinical and pathophysiological data by studying the retinal microvascularization of patients with the disease.

ELIGIBILITY:
Inclusion Criteria:

Patient Amyotrophic Lateral Sclerosis :

* Patient diagnosed with bulbar or spinal ALS defined according to El Escorial criteria (probable or certain)
* Hospitalized in a day hospital at the Angers University Hospital as part of his usual follow-up

Control subject :

* Subject not affected by the disease studied and without a history of neurological disease.
* Subject matched in age and sex to a case (patient)

For all participants:

* Major upon inclusion
* Signature of informed consent to participate in the protocol

Exclusion Criteria:

Patient Amyotrophic Lateral Sclerosis and control subject :

* Simultaneous participation in another intervention protocol with an experimental treatment
* Subject unable to express consent
* Known ophthalmologic pathology (maculopathy, glaucoma, optic neuropathy, retinopathy whatever the etiology)
* Diabetic subject
* Cardiovascular history
* Inability to perform the ophthalmological examinations of the study
* Pregnant, lactating or parturient woman
* Subject under duress psychiatric care
* Subject to legal protection
* Subject not affiliated or not beneficiary of a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2021-02-12 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Compare the angiographic optical coherence tomography examination in patients with ALS in comparison with healthy controls | at inclusion
  Compare the angiographic optical coherence tomography examination in patients with ALS in comparison with healthy controls

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Angers, Angers, France